CLINICAL TRIAL: NCT04810455
Title: An In-situ, Child-led Intervention To Promote Emotion Regulation Competence in Middle Childhood: Protocol For an Exploratory Randomised Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: Committee for Children (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #18-CFC-101
Record Dates: First submitted 2021-03-15; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Emotions
Keywords: emotion regulation; child-led intervention; in-situ intervention
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purrble -- Intervention design and logic model (Experimental): The intervention takes the form of an interactive plush toy, designed to be handed over to the child and support in-the-moment soothing; see (Theofanopoulou et al 2019, Slovak et al 2018) for the design and data from previous deployments.
  The toy is introduced to the child as an anxious creature that needs kind attention from humans. When picked up, the toy emits a frantic heartbeat that slows down if the child uses calm stroking movements. If the toy is soothed for long enough, it transitions into a purring vibration indicating a calm, content state.
  Logic model underlying the intervention:
  * Level 1: in-the-moment soothing support to children in emotional moments when they would attempt to calm down.
  * Level 2: mechanisms that facilitate long-term engagement with the intervention, building on positive subjective experience of Level 1.
  * Level 3: shift in children's ER practices and implicit beliefs about emotion, after repeated experience of Levels 1-2.
  Interventions: Other: Purrble
- Non-interactive plush toy -- active control group (Active Comparator): The investigators argue that a comparison with a non-active control-such as waiting list / treatment-as-usual (i.e., nothing)-would not allow us to distinguish the hypothesised impact on in-the-moment soothing of interactivity vs. the emergence of new family routines; and would be also open to unequal social desirability bias.
  However, from the perspective of the hypothesised logic model (Levels 1-3), it is not necessary for the active control to have exactly the same form factor as the active toy, as long as it is comparable in size, shape, and appeal. In fact, the investigators have explicitly decided not to use deactivated Purrble units as active controls due to the increased risk of unblinding, whereby the participants search for or come across Purrble online (or notice the plastic enclosure with electronics inside the toy), and assume their unit is malfunctioning.
  Interventions: Other: Active control toy

INTERVENTIONS:
Other: Purrble — The objective of this study is to evaluate the impact of having access to the Purrble intervention, compared to an active control in the form of a non-interactive plush toy, on child daily emotion regulation (primary outcome) as well as a range of secondary outcomes over a period of one month.
  The investigators hypothesise that engagement with an in-situ, 'bottom-up' emotion regulation intervention which enables in-the-moment soothing for children, will lead to measurable changes in child self-regulatory behaviours over time.
  Arms: Purrble -- Intervention design and logic model
Other: Active control toy — The selected active control toy is the Wild Republic 8'' Hedgehog animal. The selection process was guided by: the plush toy needed to have analogous size, weight, quality of materials, and at least similar (if not higher) visual appeal. The investigators also made sure to include the design characteristics our prior work suggested were important for the narrative around the toy. These were selecting a similarly stylised animal (to enable emotion projection and feelings of care), as well as no visible mouth on the toy (to prevent setting an expectation about the toy's emotional state as a mouth would imply an emotional expression). Additionally, the investigators have adapted the one-page parent-facing descriptions of the narrative that come with Purrble also for the active control unit: as such, the active control families will receive the same general narrative-without the explicit mentions of the toy interactivity-and the same suggested activities for parents.
  Arms: Non-interactive plush toy -- active control group

SUMMARY:
The aim of this study is to examine, for the first time, the efficacy of a new intervention model for child-led emotion regulation -Purrble- that could be deployed across prevention and treatment contexts.

DETAILED DESCRIPTION:
Background: Emotion regulation is a key transdiagnostic risk factor for a range of psychopathologies, making it a prime target for both prevention and treatment interventions in childhood. Existing interventions predominantly rely on workshop or in-person therapy-based approaches, limiting the ability to promote emotion regulation competence for children in everyday settings and at scale. Purrble is a newly developed, inexpensive socially assistive robot-in the form of an interactive plush toy-which uses haptic feedback to support in-the-moment emotion regulation. It is accessible to children as needed in their daily lives, without the requirement for a priori training. While qualitative data from prior studies show high engagement in-situ and anecdotal evidence of the robot being incorporated into children's emotion regulation routines, there is so far no quantitative evidence of the intervention's impact on child outcomes.

Objective: The aim of this study is to examine, for the first time, the efficacy of a new intervention model for child-led emotion regulation-Purrble-that could be deployed across prevention and treatment contexts.

Methods: A total of 120 children aged 8-10 will be selected from an 'enriched' non-clinical US population: for inclusion, the cutoff for parent's rating of child dysregulation will be 10 points or higher on the total difficulties score on the Strengths and Difficulties Questionnaire. This cutoff selects for a measurable-but not necessarily clinical-level of the child's emotion regulatory difficulties. The selected families will be randomly assigned with .5 probability to receive either Purrble or an active control (non-interactive plush toy). The primary outcome will be a daily EMA measure of child emotion regulation capability (as reported by parents) over a period of 4 weeks. Exploratory analysis will investigate the intervention impact on secondary outcomes of child emotion regulation, collected weekly over the same 4 week period, with follow-ups at 1 month and 6 months post-deployment. Quantitative data will be analysed on an intent-to-treat basis. A proportion of families (~30% of the sample) will be interviewed post-deployment as part of process analysis.

ELIGIBILITY:
Inclusion Criteria:

* child aged 8-10
* parent-reported score of 10 or higher for the total difficulties score on the Strength and Difficulties (SDQ) questionnaire

Exclusion Criteria:

* child participating in another mental health intervention
* parent and/or child not fluent in English (as all measurement scales are in English)

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-03-13 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Perceived child emotion regulation ability | Daily, for the 4-week long deployment period
  Composite end-of-day 4-item parent-report measure of the perceived child emotion regulation ability throughout the day. The composite score for each day will be computed as the mean value across the 4 items:
  * Today, to what extent was the participant's child able to take difficult things in stride?
  * Today, to what extent did the participant's child get easily triggered or upset?
  * Today, to what extent was the participant's child able to calm down easily if upset?
  * Today, to what extent did the participant's child get very emotional even after the littlest things?
  These items were selected as tapping into the proximal emotion regulation behaviour that (a) would be affected if the intervention is effective, (b) directly observable by parents, (c) state-based to enable daily measurement, (d) connected to the intervention theory of change.

SECONDARY OUTCOMES:
Daily parent-report EMA -- child daily mood (mDES) | Daily, for the 4-week long deployment period
  Measured by selected mDES (Fredrickson et al 2003) emotion triplets, balancing 2 negative and 2 positive sets, whilst being informed by prior qualitative studies. The items are listed below, all measured on a visual analogue scale with not at all and extremely as the anchors.
Daily parent-report EMA -- daily engagement | Daily, for the 4-week long deployment period
  Daily engagement item asks about general perception of engagement with the toy ("How much did the participant's child play with the toy today?", measured on a visual analogue scale with <not even once> and <they were inseparable> as the anchors).
Daily parent-report EMA -- reaction to triggering events | Daily, for the 4-week long deployment period
  Series of explorative items examining the child's reaction after potentially triggering events. The investigators will first ask the parents "Did anything happen today that would typically upset the participant's child?". The purpose of these items to gain qualitative understanding of the toys' use around challenging situations and to guide post-deployment interviews.
Weekly questionnaires for parents -- child emotion regulation (SDQ) | at baseline (just before intervention/control toys are delivered); and then weekly for a period of one month (end of week 1, week 2, week 3, week 4); and then at 1-month and 6-month follow-up.
  These include parent reports on distal outcomes of parent-reported emotional and behavioural difficulties of the child will be measured by the 25-item Strength and Difficulties Questionnaire (SDQ).
Weekly questionnaires for parents -- child emotion regulation (ERC) | at baseline (just before intervention/control toys are delivered); and then weekly for a period of one month (end of week 1, week 2, week 3, week 4); and then at 1-month and 6-month follow-up.
  These include parent reports on distal outcomes of parent-reported emotion regulation lability and competence will be measured by the 24-item Emotion Regulation Checklist (ERC) questionnaire.
Weekly questionnaires for parents -- engagement (TWEETS) | weekly for a period of one month (end of week 1, week 2, week 3, week 4); and then at 1-month and 6-month follow-up.
  Parent-reported behavioural, cognitive, and affective engagement with the intervention will be measured by an adapted version of the TWEETS questionnaire, a new, promising instrument specifically designed to measure engagement with digital mental health interventions, with good reliability in prior studies.
Weekly questionnaires for children (DERS) | 5 data points collected: at baseline, and end of week 1, week 2, week 3 and week 4
  Child-reported emotion dysregulation will be measured by a shortened version of Brief Difficulties in Emotion Regulation Scale (DERS), following prior work with children of similar ages (Schneider et al 2020). DERS has been developed to measure clinically relevant difficulties in emotion regulation, across 6 factor-analytically-derived subscales. The DERS questionnaire has been used extensively to facilitate understanding of how emotion dysregulation is associated with psychiatric symptoms, and to measure treatment progress.
Weekly questionnaires for children (ER beliefs) | 5 data points collected: at baseline, and end of week 1, week 2, week 3 and week 4
  Child-reported beliefs about emotion regulation will be measured by an adapted ER beliefs questionnaire (Ford et al 2017), asking children to pick one out of four statements (e.g., "I cannot control my feelings at all"; "I can control my feelings a little"; "I can control my feelings a lot"; I can control my feelings all the time") rather using the original Likert scale statements asking about agreement.

OTHER OUTCOMES:
Post-deployment interviews (process analysis) | One time, within 2 weeks following the primary data collection period
  The investigators will collect semi-structured interview data with parents of up to 40% of the experimental group sample (20-25 families), and approximately 25% or the control group (15 families).
  The investigators will be specifically aiming to recruit families who show the highest / lowest change in the outcome data over the primary period to qualitatively understand the potential moderators of intervention response for future research.
  The semistructured interview guide will explore the engagement with the toy; any qualitative changes in child or family behaviour patterns that parents notice; appropriation (i.e., how the intervention ended up being used by different participants), and use trajectory over time.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slovak P, Ford BQ, Widen S, Dauden Roquet C, Theofanopoulou N, Gross JJ, Hankin B, Klasnja P. An In Situ, Child-Led Intervention to Promote Emotion Regulation Competence in Middle Childhood: Protocol for an Exploratory Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 9;10(11):e28914. doi: 10.2196/28914. PMID 34751666